CLINICAL TRIAL: NCT05582239
Title: Measure of Vaccine Effectiveness to Prevent Hospitalizations for Viral Respiratory Infections in Adults
Acronym: RESPIVAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: P95 (Industry); I-REIVAC (Unknown); EPICONCEPT (Unknown); Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS0285s
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Severe Acute Respiratory Infection (SARI); Influenza; COVID-19
Keywords: Severe acute respiratory infection (SARI); Vaccine effectiveness; Influenza; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Swab respiratory samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, multicentric, observational test negative design study on adults hospitalized for Severe Acute Respiratory Infection (SARI), regardless of their vaccination status.

DETAILED DESCRIPTION:
Participation to the study will be systematically proposed to all patients hospitalized fitting inclusion criteria. Patient's screening will be done in emergency department or hospital department with direct admission. Medical investigators explain the objectives of the studies, procedure and propose the patient to participate in the study. Socio-demographic data, clinical and virological data will be collected in an electronic clinical research form.

A follow-up at 1 and 3 months after hospitalization discharge will be scheduled to evaluate health status.

The remainder of respiratory samples that have been performed for care will be used for further testing depending on epidemiological situation and will be stored at -80°C.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Admitted in a hospital for at least 24 h
* Presents SARI criteria within onset within the last 14 days before sampling and less than 48 h after hospitalisations:

At least one of the following signs (without treatment): fever or feverishness, malaise, headache, myalgia or sign of fatigue (loss of weight or anorexia or confusion or dizziness) Associated with at least one respiratory symptom or sign (cough, sore throat or shortness of breath; or tachypnoea or signs of low oxygen saturation)

* completed non-opposition form
* Respiratory samples within 14 days after symptoms onset, in the context of care

Exclusion Criteria:

* Contraindication of vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients presenting with SARI symptom onset in the first 14 days
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Vaccine effectiveness | up to 48 hours
  Comparison of the number of virologically confirmed cases of vaccine preventable Severe Acute Respiratory Infections (SARI) among hospitalized vaccinated patients compared with unvaccinated patients.

SECONDARY OUTCOMES:
Covid-19 vaccine effectiveness | up to 48 hours
  Comparison of numbers of hospitalized cases with documented COVID-19 infection in vaccinated and unvaccinated patients according to:
  * Age
  * comorbidities
  * Vaccine schedule (numbers of doses and brand)
  * date of vaccination
  * SARS-CoV-2 Variant
Influenza vaccine effectiveness | up to 48 hours
  Comparison of numbers of hospitalized cases with documented flu in vaccinated and unvaccinated according to:
  * Age
  * Comorbidities
  * Vaccine brand
  * Date of vaccination
  * Previous vaccination
  * Viral strain
Prevalence of viral and bacterial co-infections | up to 48 hours
  Prevalence of other viruses and bacteria detected by PCR, antigen tests, microbiology samples.
Incidence of SARI by site | up to 12 months
  Incidence rate of SARI by sites
Clinical burden of SARI | up to 3 months
  European Quality of Life by 5 Dimension (EQ5D) score assessed at 1 month and 3 months after hospitalization discharge. Scale from 0 to 100 with 0 corresponding to the worst quality of life.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU, Dijon
  - Groupement hospitalier Edouard Herriot, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - CHU, Nantes
  - Hôpital Cochin, Paris
  - Hôpital Bichat, Paris
  - CHU, Rennes
  - CHU, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No